CLINICAL TRIAL: NCT05829850
Title: An Effectiveness and Safety 6 Months Study of 3 Injections One Week Apart of SYNOLIS VA 40/80 in the Treatment of Symptomatic Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aptissen SA (Industry)
Collaborators: Noblewell (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMCF2ML Multishot
Record Dates: First submitted 2023-03-21; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Osteo Arthritis Knee
Keywords: Osteoarthritis; Knee Osteoarthritis; Hyaluronic acid
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SYNOLIS VA 40/80 (Experimental): SYNOLIS VA 40/80 (hyaluronic acid 40 mg, sorbitol 80 mg), intra-articular injection
  Interventions: Device: SYNOLIS VA 40/80

INTERVENTIONS:
Device: SYNOLIS VA 40/80 — Three 2mL injections of SYNOLIS VA 40/80, one week apart

SUMMARY:
Multicentre, independent assessment study on SYNOLIS VA 40/80 over a period of 24 weeks

ELIGIBILITY:
Inclusion Criteria:

* Patient between 35 and 75 years old
* Patients with knee osteoarthritis. The diagnosis is based on the following American College of Rheumatology (ACR) classification:

  * Knee pain
  * Positive radiography (presence of osteophytes)
  * Morning stiffness < 30 min and/or crepitus while walking
* Symptoms related to knee osteoarthritis for at least 6 months
* Treatment failure (i.e. ineffective response) with analgesics and/or NSAIDs or intolerance to NSAIDs or low-grade opioids
* Kellgren-Lawrence radiographic stage: I - III (pre-inclusion radiography)
* VAS pain index score ≥ 40 mm (VAS 0-100 mm) on the knee to be treated
* Contralateral knee pain < 10 mm (VAS) compared to treated knee
* Patient signed inform consent form

Exclusion Criteria:

* Inability to understand the study or language used to be informed/sign the consent
* Participation in another clinical trial within 4 weeks prior to the start of the trial, and commitment to non-participation within 4 weeks following the end of the trial
* Intraarticular injection of hyaluronic acid in target knee within the 6 months prior to inclusion
* Patient who has received an intra-articular (IA) or intra-muscular (IM) steroid injection within the 3 months prior to inclusion or has taken oral corticosteroids within the month prior to inclusion
* Joint, bone, ligament, or any local or loco-regional surgery of the leg involved, arthroscopic operation on the target knee within the 3 months prior to inclusion
* Any recent trauma to the leg involved, including a sprain, dislocation within the 3 months prior to inclusion
* Rheumatoid arthritis, joint condition or any other inflammation and arthritis
* Lupus
* Dermatological disorder or any epidermal conditions that prevent an intraarticular injection
* Visible remarkable joint effusion of the target knee during physical examination evidenced by a protuberance or positive ballottement of the patella
* Evidence of a subchondral fracture, meniscal lesion, presence of bone or cartilage fragments, horizontal meniscal lesion tear (FLAP) in the target knee
* Osteonecrosis (1 or both knees)
* Daily dosage > 101 mg of acetylsalicylic acid as part of cardiovascular preventive treatment (antithrombotic). If dose < 101 mg, must be maintained during the study
* Known intolerance/hypersensitivity/allergy to any of the components in either product, SYNOLIS VA
* Fibromyalgia
* Patient of childbearing potential, pregnant or breast-feeding known at inclusion or in the planning phase during the study unless willing to use contraceptives through the whole duration of the study
* Excessive and repeated consumption of alcohol or illicit substances
* Any medical condition that may interfere with the proper conduct of the study (including any surgery or hospitalisation)

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Difference in total Western Ontario and McMaster Universities Arthritis index (WOMAC) score total between D168 and inclusion visit. | 168 days
  The Western Ontario and McMaster Universities Arthritis index (WOMAC) is a 24-item, condition-specific questionnaire available in a 5-point Likert and 100 mm visual analog scale (VAS) as well as an 11-box numerical rating scale, composed of three subscales: pain (5 questions), stiffness (2 questions) and physical function (17 questions). VAS was used in this study, with a score of 0 for no pain and 100 mm for the worst pain one can image)

SECONDARY OUTCOMES:
Change in pain measurements, assessed using the Western Ontario and McMaster Universities Arthritis (WOMAC) pain severity index, as compared to D0 | up to 168 days
  The Western Ontario and McMaster Universities Arthritis index (WOMAC) is a 24-item, condition-specific questionnaire available in a 5-point Likert and 100 mm visual analog scale (VAS) as well as an 11-box numerical rating scale, composed of three subscales: pain (5 questions), stiffness (2 questions) and physical function (17 questions). VAS was used in this study, with a score of 0 for no pain and 100 mm for the worst pain one can image)
Change in the Western Ontario and McMaster Universities Arthritis (WOMAC) functional severity index, as compared to D0 | up to 168 days
  The Western Ontario and McMaster Universities Arthritis index (WOMAC) is a 24-item, condition-specific questionnaire available in a 5-point Likert and 100 mm visual analog scale (VAS) as well as an 11-box numerical rating scale, composed of three subscales: pain (5 questions), stiffness (2 questions) and physical function (17 questions). VAS was used in this study, with a score of 0 for no pain and 100 mm for the worst pain one can image)
Change in the Western Ontario and McMaster Universities Arthritis (WOMAC) stiffness severity index, as compared to D0 | up to 168 days
  The Western Ontario and McMaster Universities Arthritis index (WOMAC) is a 24-item, condition-specific questionnaire available in a 5-point Likert and 100 mm visual analog scale (VAS) as well as an 11-box numerical rating scale, composed of three subscales: pain (5 questions), stiffness (2 questions) and physical function (17 questions). VAS was used in this study, with a score of 0 for no pain and 100 mm for the worst pain one can image)
Pain at walking on a 100 mm VAS | up to 168 days
Percentage of subjects using analgesics | up to 168 days
  New NSAID / analgesics drugs usage
Measurement of relief satisfaction by the patient | 168 days
  7-point Likert scale (1 point very unsatisfied to 7 points for very satisfied)
Measurement of therapeutic efficacy by the investigator (assessor) | 168 days
  7-point Likert scale (1 point very unsatisfied to 7 points for very satisfied)

OTHER OUTCOMES:
Safety and tolerability of SYNOLIS VA 40/80 assessed with adverse events monitoring throughout the study duration | 168 days

CONTACTS AND LOCATIONS:
Locations (3):
- Poland (3):
  - SPORTO oddzial na ulicy Miedzianej, Lodz
  - SPORTO oddzial na ulicy Książka (2nd site location), Lodz
  - Carolina Medical Center, Warsaw